CLINICAL TRIAL: NCT01306448
Title: Safety Evaluation of the Vibrating Capsule in Aiding Reliving Constipated Individuals
Brief Title: Safety Evaluation of the Vibrating Capsule
Acronym: Vibrant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrant Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vibrant-09-MS-CTIL
Record Dates: First submitted 2011-02-21; First posted 2011-03-01 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Constipation
Keywords: constipation; gastro; vibrating capsule; safety
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vibrating capsule (Experimental)
  Interventions: Device: Vibrant capsule

INTERVENTIONS:
Device: Vibrant capsule — vibrating capsule
  Other Names: Vibrant

SUMMARY:
The study will assess the safety of the vibrating capsule in healthy volunteers first and than for constipation relief constipated individuals.

DETAILED DESCRIPTION:
Healthy volunteers will be followed for safety for 7 days after taking the capsule.

Constipated individuals will be first followed for 2 weeks and than they will use the capsule for 7.5 weeks period. Safety and efficacy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-60 years
* Ability of subject to understand character and individual consequences of clinical trial
* Written informed consent must be available before enrollment in the trial
* For women with childbearing potential, adequate contraception

Exclusion Criteria:

* Patient with Diverticulosis
* Patient must not use protocol-defined prohibited medicine
* History of or current diagnosis of cardiovascular ischemic disease (e.g., angina pectoris, myocardial infarction, transient ischemic attack or stroke and including findings suggestive of ischemia on an ECG such as changes in ST segment and T waves, and / or Q wave)
* Clinical evidence of significant (as judged by the Investigator) respiratory, cardiovascular, renal, hepatic-biliary, endocrine, psychiatric or neurologic diseases or presence of abdominal adhesions
* Presents of pacemakers
* History of or current eating disorder such as anorexia or bulimia or compulsory overeating.
* Diagnosis of mega-rectum or colon, a history of intestinal obstruction, congenital anorectal malformation, clinically significant rectocele, or any evidence of intestinal structural abnormality including gastrointestinal resection that affected bowel transit or any evidence of intestinal carcinoma, of inflammatory bowel disease or of alarm symptoms such as weight loss, rectal bleeding, or anemia.
* Actively participating in another clinical trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 7.5 weeks of treatment period
  Safety will be assessed descriptively by summarizing AEs, clinical laboratory test results, vital sign measurements, and ECG measurements

SECONDARY OUTCOMES:
Change in spontaneous bowel movement per week compared to baseline | 9.5 weeks
  Efficacy will be assessed by increase of more than one complete spontaneous bowel movement per week during the 7.5 weeks of treatment compared to 2 weeks baseline
Patient assessment of capsule tolerability | 7.5 weeks of treatment period
  Comfort and tolerability will be assessed by the patient. Tolerability evaluation will include: assessment of bowel habits, constipation, distention/bloating, abdominal discomfort/pain, patients assessment of impact of constipation on quality of life.

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Tel Aviv Souraski medical Center, Tel Aviv, Israel
  - Barzilai MC, Ashkelon
  - Italian Hospital, Nazeret